CLINICAL TRIAL: NCT02364986
Title: Immune- and miRNA-response to Recombinant Interferon Beta in Healthy Volunteers and Patients With Relapsing Remitting Multiple Sclerosis
Acronym: RESI
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: PD Dr. Marcus Müller (Other)
Collaborators: BfARM, Bonn (Unknown); DZNE, Bonn (Unknown)
Responsible Party: Sponsor-Investigator, PD Dr. Marcus Müller, PD Dr. Marcus M Müller, University Hospital, Bonn
Organization: University Hospital, Bonn (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEU-201201-RESI
Record Dates: First submitted 2014-12-10; First posted 2015-02-18 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-06

CONDITIONS: Relapsing-remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Interferon beta-1a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rebif/Avonex (Experimental): Rebif® 44µg (day 1, 3, 5 and 8) s.c. Avonex 30µg (day 1 and 8) i.m.
  Interventions: Drug: Rebif®; Drug: Avonex

INTERVENTIONS:
Drug: Rebif® — Rebif® 44µg (day 1, 3, 5 and 8) s.c.
  Other Names: Interferon beta 1a
Drug: Avonex — Avonex 30µg (day 1 and 8) i.m.
  Other Names: Interferon beta 1a

SUMMARY:
There are two standard and a few second line treatments for RRMS. Since the disease cannot be cured by these existing treatments and all treatment options have significant limitations, there is the need to develop new treatment strategies to improve therapy of patients with RRMS. We developed a RIG-I ligand as a new therapeutic strategy for patients with MS. The RIG-I ligand functions partially via induction of Interferon beta (IFN-b), but has advantages over therapy with recombinant IFN-b. Identification of suitable biomarkers to monitor treatment with RIG-I ligand and to guide the dose steps would help to increase the safety of the volunteers in the early clinical trials with RIG-I ligand.

The RESI study is designed to analyse immune readouts and potential biomarkers such as type I IFN levels, type I IFN dependent immune activation and miRNA expression following Rebif or Avonex (Interferon beta 1a) application. Rebif is applied s.c. at a dose of 44 µg three times a week (on day 1,3,5 and 8), and Avonex i.m. at a dose of 30µg once a week (on day 1 and 8), as they are routinely used in RRMS-therapy. The immune readouts are assessed on day 1, 3, 5 and 8 immediately before application of Rebif/Avonex and on day 1 and 8 at 1 / 6 / 12 /24 hrs after Rebif/Avonex application by analysing blood samples. Since studies of the RIG-I ligand will start in healthy volunteers and will be continued in MS patients we need data from both populations since they could show significant differences in response to IFN-b. Thus, the RESI study includes healthy volunteers, RRMS-patients already under Rebif/Avonex treatment, and RRMS-patients who have to yet started a therapy with Rebif/Avonex.

DETAILED DESCRIPTION:
Study subjects receive either Rebif or Avonex. Rebif is applied s.c. at a dose of 44 µg on day 1, day 3, day 5 and day 8, Avonex i.m. at a dose of 30µg on day 1 and 8. Blood samples are taken before application and on day 1 and 8 at 1 / 6 / 12 /24 hrs after Rebif/Avonex application to analyse the occuring immune response. The total duration of the trial for the individual subject are 9 days. An MRI ist performed before the first application of IMP and at the end of the study to investigate the correlation of Rebif/Avonex application and depression.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation in this study as proven by written informed consent
* Female or male patients with relapsing remitting MS according to McDon-ald-criteria (2010 revision) and decision for IFN-b treatment according to routine clinical criteria (not applying for healthy volunteers)
* Expanded Disability Status Scale (EDSS) between 0.0 and 6.0 (not applying for healthy volunteers)
* Naïve for IFN-b therapy (not applying for RRMS patients already under treatment)
* Age between 18 and 65 years
* Ability to follow study instructions and likely to attend and complete all required visits
* Adequate organ function as described below:

  * Adequate bone marrow reserve:

    * White blood cell (WBC) count ≥ 3000/µl,
    * granulocyte count > 1500/µl,
    * platelets ≥ 100000/µl,
    * haemoglobin ≥ 10 g/dl
  * Adequate liver function

    * bilirubin < 1.5 times above upper limit of normal range (ULN) (the higher concentrations are only allowed for patients with RRMS)
    * alanine transaminase (ALT/SGPT) and aspartate transaminase (AST/SGOT) < 3 times ULN (the higher concentrations are only allowed for patients with RRMS)
  * Adequate renal function: creatinine < 1.5 times ULN (the higher concentrations are only allowed for patients with RRMS)
  * TSH within normal limits
  * Adequate blood clotting:

    * INR and PTT within normal limits
* Male and female patients with reproductive potential must use an approved contraceptive method during and for 3 months after the trial (Pearl index <1; Oral hormonal contraception must be used in combination with a barrier device due to elevated risk of nausea. Use of an intrauterine device made of copper is not allowed for healthy volunteers due to MRI)
* Pre-menopausal female patients with childbearing potential: a negative serum pregnancy test must be obtained prior to treatment start
* MRI study: only healthy participants

Exclusion Criteria:

* Subjects not able to give consent
* Subject without legal capacity who is unable to understand the nature, scope, significance and consequences of this clinical trial
* Patients suffering from a form other than relapsing remitting Multiple Sclerosis (not applying for healthy volunteers)
* Patients with a MS relapse within 30 days before study inclusion
* EDSS >6.0 (not applying for healthy volunteers)
* Patients with known allergy or hypersensitivity to Interferon-beta or ingredients of the injection solution
* Subjects with a physical or psychiatric condition/ a systemic disease which at the investigator's discretion may compromise safety of the subject, may confound the trial results, may interfere with the subject's participation in this clinical trial or may prevent sufficient compliance
* Known or persistent abuse of medication, drugs or alcohol
* Prior malignancy (unless adequately treated carcinoma in situ of the cervix or nonmelanoma skin cancer). If prior malignancy was diagnosed and definitively treated at least 5 years previously with no subsequent evidence of recurrence the subject can be enrolled at the discretion of the investigator
* Prior chemotherapy, systemic or local treatment with DNA-damaging and immune-modulating agents, tyrosine kinase inhibitors or anti-angiogenic agents for any cancer
* History of major depression, suicide attempt in the past, ongoing suicidal thoughts
* Cardiac insufficiency (NYHA III or IV), cardiomyopathy, significant cardiac dysrhythmia, unstable or advanced ischemic heart disease, or significant hypertension at rest (BP > 180/110 mmHg)
* HIV, Hepatitis B or C infection or any relevant infectious disease which might interfere with the study procedures and results (at the discretion of the investigator)
* Women who are pregnant or breast-feeding
* Comedication with corticosteroids
* Female Patients with reproductive potential who do not accept to use contraception during the trial and 3 months thereafter
* Treatment in another clinical trial with therapeutic intervention or use of any other investigational medicinal product (IMP) during the trial or within the 30 days but at least 5 times the half life of the IMP before enrolment
* Very poor peripheral veins and pronounced fear of blood drawings
* Patients with history of epileptic seizures and / or under medical therapy with antiepileptic drugs
* MRI study: Metal implants (eg pacemaker, inner-ear prosthesis, nerve stimulator, implanted defibrillator, infusion pump, artificial joints), wearing of magnetic or metallic objects that cannot be removed from the body (such as body piercing, dental prosthesis, implanted electrodes, contraceptive coil, acupuncture needle), tattoos & permanent makeup, claustrophobia, tinnitus, inability to lie on the back for an extended period of time, previous surgery on heart or head

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Change of mRNA (IFN-b, CXCL10, IL-6, MxA and 5'-3'OAS) and protein expression (IFN-b, CXCL10, IL-6) in peripheral blood mononuclear cells/ serum | before / after 1hr / 6 hrs / 12 hrs / 24 hrs
  PBMCs and Serum are isolated from the blood before and at different time points after the application of Rebif/Avonex on day 1, 3, 5, and 8 (before / after 1hr / 6 hrs / 12 hrs / 24 hrs) to assess the changes in mRNA and protein expression related to Rebif/Avonex administration

SECONDARY OUTCOMES:
Change of mRNA and miRNA expression in peripheral blood mononuclear cells and serum in healthy volunteers as well as in patients with RRMS | before / after 1hr / 6 hrs / 12 hrs / 24 hrs
  PBMCs and Serum are isolated from the blood before and at different time points after the application of Rebif/Avonex on day 1,3,5, and 8 (before / after 1hr / 6 hrs / 12 hrs / 24 hrs) to assess the change in mRNA and miRNA expression determined by Chip Array related to Rebif/Avonex administration
Correlation of Rebif/Avonex side effects in patients with RRMS and healthy volunteers with changes in IFN-b, CXCL10, MxA, 5'-3'OAS, IL-6 serum levels, gene- and miRNA expression pattern and functional immune tests | day 1 (+1 hr / 6hrs /12 hrs after 1. Rebif/Avonex application)
  Rebif/Avonex side effects and the occuring immune response (measured by protein- / gene- / miRNA-levels from PBMCs and Serum) are correlated at different time points after the application of Rebif/Avonex on day 1,3,5, and 8 (before / after 1hr / 6 hrs / 12 hrs / 24 hrs)
Correlation of Rebif/Avonex side effects in patients with RRMS and healthy volunteers with changes in IFN-b, CXCL10, MxA, 5'-3'OAS, IL-6 serum levels, gene- and miRNA expression pattern and functional immune tests | day 2 (24 hrs after 1.Rebif/Avonex application)
  Rebif/Avonex side effects and the occuring immune response (measured by protein- / gene- / miRNA-levels from PBMCs and Serum) are correlated at different time points after the application of Rebif/Avonex on day 1,3,5, and 8 (before / after 1hr / 6 hrs / 12 hrs / 24 hrs)
Correlation of Rebif/Avonex side effects in patients with RRMS and healthy volunteers with changes in IFN-b, CXCL10, MxA, 5'-3'OAS, IL-6 serum levels, gene- and miRNA expression pattern and functional immune tests | day 3 (48 hrs after 1.Rebif/Avonex application)
  Rebif/Avonex side effects and the occuring immune response (measured by protein- / gene- / miRNA-levels from PBMCs and Serum) are correlated at different time points after the application of Rebif/Avonex on day 1,3,5, and 8 (before / after 1hr / 6 hrs / 12 hrs / 24 hrs)
Correlation of Rebif/Avonex side effects in patients with RRMS and healthy volunteers with changes in IFN-b, CXCL10, MxA, 5'-3'OAS, IL-6 serum levels, gene- and miRNA expression pattern and functional immune tests | day 5 (48 hrs after 2.Rebif/ 96 hrs after 1. Avonex application)
  Rebif/Avonex side effects and the occuring immune response (measured by protein- / gene- / miRNA-levels from PBMCs and Serum) are correlated at different time points after the application of Rebif/Avonex on day 1,3,5, and 8 (before / after 1hr / 6 hrs / 12 hrs / 24 hrs)
Correlation of Rebif/Avonex side effects in patients with RRMS and healthy volunteers with changes in IFN-b, CXCL10, MxA, 5'-3'OAS, IL-6 serum levels, gene- and miRNA expression pattern and functional immune tests | day 8 (72 hrs after 3. Rebif application, +1 hr / 6hrs /12 hrs after 4. Rebif/ 2. Avonex application)
  Rebif/Avonex side effects and the occuring immune response (measured by protein- / gene- / miRNA-levels from PBMCs and Serum) are correlated at different time points after the application of Rebif/Avonex on day 1,3,5, and 8 (before / after 1hr / 6 hrs / 12 hrs / 24 hrs)
Correlation of Rebif/Avonex side effects in patients with RRMS and healthy volunteers with changes in IFN-b, CXCL10, MxA, 5'-3'OAS, IL-6 serum levels, gene- and miRNA expression pattern and functional immune tests | day 9 (24 hrs after 4. Rebif/ 2. Avonex application)
  Rebif/Avonex side effects and the occuring immune response (measured by protein- / gene- / miRNA-levels from PBMCs and Serum) are correlated at different time points after the application of Rebif/Avonex on day 1,3,5, and 8 (before / after 1hr / 6 hrs / 12 hrs / 24 hrs)
Psychometric testing: correlation between Rebif/Avonex administration and scores in depression and anxiety scales | before / day 9
  Psychometric tests are performed before the first application of Rebif/Avonex and at the end of the study at day 9 (24 hrs after 4.Rebif application) and changes between the 2 time points are evaluated
MRI: Changes in regional cerebral blood flow at rest (arterial spin labeling) and their correlation with psychometric outcome variables and with transcriptome data | before / day 9
  MRI is performed before the first application of Rebif/Avonex and at the end of the study at day 9 (24 hrs after 4.Rebif application) and changes between the 2 time points are evaluated
Changes in functional neuroimaging endophenotypes in the limbic system or prefrontal cortex that constitute possible markers of anxiety and depression and their correlation with psychometric outcome variables | before / day 9
  Neuroimaging endophenotypes are assessed before the first application of Rebif/Avonex and at the end of the study at day 9 (24 hrs after 4.Rebif/ 2. Avonex application) and changes between the 2 time points are evaluated
Changes of IFN-b, CXCL10, MxA, 5'-3'OAS, IL-6 serum levels, gene- and miRNA-expression pattern and functional immune tests between healthy volunteers, RRMS-patients naïve to IFN-b and RRMS-patients with established IFN-b treatment | before / after 1hr / 6 hrs / 12 hrs / 24 hrs
  PBMCs and Serum are isolated from the blood before and at different time points after the application of Rebif/Avonex on day 1, 3, 5 and 8 (before / after 1hr / 6 hrs / 12 hrs / 24 hrs) to assess the changes in protein- / gene- and miRNA expression related to Rebif administration

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Müller, PD Dr., Principal Investigator — Department of Neurology University Hospital Bonn
Locations (2):
- Germany (2):
  - Department of Neurology, Bonn
  - Phase I Unit, Bonn

REFERENCES:
- [Derived] Coenen M, Hinze AV, Mengel M, Fuhrmann C, Ludenbach B, Zimmermann J, Dykstra V, Fimmers R, Viviani R, Stingl J, Holdenrieder S, Muller M, Hartmann G, Coch C. Immune- and miRNA-response to recombinant interferon beta-1a: a biomarker evaluation study to guide the development of novel type I interferon- based therapies. BMC Pharmacol Toxicol. 2015 Sep 22;16:25. doi: 10.1186/s40360-015-0025-x. PMID 26392348